CLINICAL TRIAL: NCT01981954
Title: A Phase 3, Open-Label, Baseline-controlled, Multi-center, Sequential Dose-Titration Study to Assess the Pharmacokinetics, Long-Term Efficacy and Safety of Solifenacin Succinate Suspension in Children From 6 Months to Less Than 5 Years of Age With Neurogenic Detrusor Overactivity
Brief Title: A Clinical Study to Investigate How Solifenacin Fluid is Taken up, How Long it Stays in the Body and How Effective and Safe it is in Treating Children Aged From 6 Months to Less Than 5 Years With Symptoms of Neurogenic Detrusor Overactivity (NDO)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Europe B.V. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 905-CL-074; 2012-003178-22 (EudraCT Number)
Record Dates: First submitted 2013-11-06; First posted 2013-11-13 (Estimated); Results first posted 2018-06-21 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Neurogenic Detrusor Overactivity; Pediatric
Keywords: Solifenacin succinate suspension; Efficacy; Safety
MeSH Terms: interventions — Solifenacin Succinate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Solifenacin succinate (Experimental): Children aged 6 months to less than 5 years were treated with sequential titrated doses of solifenacin up to 12 weeks in the Titration period after which a fixed dose of solifenacin was given for at least 40 weeks in the Fixed-dose assessment period. Children received solifenacin once daily during these 2 periods.
  Interventions: Drug: Solifenacin succinate

INTERVENTIONS:
Drug: Solifenacin succinate — Oral suspension
  Other Names: solifenacin; YM905; solifenacin succinate suspension

SUMMARY:
The purpose of this study was to evaluate long term efficacy and safety of treatment with solifenacin succinate (the study drug) in children with neurogenic detrusor overactivity after multiple dose administration.

DETAILED DESCRIPTION:
In some children with a severe form of spina bifida (which is the consequence of a spinal cord defect), the bladder muscle (detrusor) contracts strongly and without warning (also known as neurogenic detrusor overactivity) and the urethra (the passage connecting the bladder with outside) does not relax. Though these children cannot void, urine leakage can happen when the overactive contractions are strong, and/or the pressure in the bladder is so high that it overcomes the closed urethra (overflow at high filling bladder pressure). This high bladder pressure puts these children at risk for kidney damage and can decrease the quality of the bladder. Therapy was aimed to decrease the high filling bladder pressure and the overactive detrusor contractions.

ELIGIBILITY:
Inclusion Criteria:

* Myelomeningocoele
* Documented diagnosis of NDO, confirmed by urodynamics
* DSD (detrusor sphincter dyssynergia)
* Practicing clean intermittent catheterization (CIC)

Exclusion Criteria:

* Know genitourinary condition (other than NDO) that may cause incontinence
* Bladder augmentation surgery
* Current faecal impaction
* Electro-stimulation therapy within 2 weeks prior to visit
* Subjects with the following gastro-intestinal problems: partial or complete obstructions, decreased motility like paralytic ileus, subjects at risk of gastric retention
* Reflux grade 3 to 5
* Current urinary tract infection

Ages: 6 Months to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 23 (Actual)
Dates: Start 2013-09-25 (Actual); Primary Completion 2015-12-18 (Actual); Study Completion 2015-12-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Europe B.V.
Locations (8):
- Site US1008 Pediatric Urology Associates, P.C., Tarrytown, New York, United States
- Site BE3203 Gent University Hospital, Ghent, Belgium
- Site PH6301 Philippines Children's Medical Center, Manila, Philippines
- Poland (2):
  - Site PL4803 Uniwersyteckie Centrum Kliniczne, Gdansk
  - Site PL4801 Pomnik-Centrum Zdrowia Dziecka, Warsaw
- South Korea (2):
  - Site KR8207 Seoul National University Hospital, Seoul
  - Site KR8201 Severance Hospital, Seoul
- Site GB4401 Sheffield Children's Hospital, Sheffield, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- [Derived] Tannenbaum S, den Adel M, Krauwinkel W, Meijer J, Hollestein-Havelaar A, Verheggen F, Newgreen D. Pharmacokinetics of solifenacin in pediatric populations with overactive bladder or neurogenic detrusor overactivity. Pharmacol Res Perspect. 2020 Dec;8(6):e00684. doi: 10.1002/prp2.684. PMID 33231929
- [Derived] Franco I, Hoebeke P, Baka-Ostrowska M, Bolong D, Davies LN, Dahler E, Snijder R, Stroosma O, Verheggen F, Newgreen D, Bosman B, Vande Walle J. Long-term efficacy and safety of solifenacin in pediatric patients aged 6 months to 18 years with neurogenic detrusor overactivity: results from two phase 3 prospective open-label studies. J Pediatr Urol. 2020 Apr;16(2):180.e1-180.e8. doi: 10.1016/j.jpurol.2019.12.012. Epub 2019 Dec 27. PMID 32007426
- See also: Link to results on the Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=242

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Children aged 6 months to < 5 years old with neurogenic detrusor overactivity (NDO) were enrolled from Belgium (1 site), United Kingdom (1 site), Poland (2 sites), United States (1 site), the Philippines (1 site) and South Korea (2 sites).
Pre-assignment Details: Children who met the eligibility criteria were treated with sequential doses of solifenacin up to 12 weeks to determine each participant's optimal dose, after which a fixed dose of solifenacin was given for at least 40 weeks. A washout period was required between screening and baseline if the children were being treated with antimuscarinic agents.
Groups:
- Solifenacin Succinate: Children aged 6 months to < 5 years were treated with sequential titrated doses of solifenacin up to 12 weeks in the Titration period after which a fixed dose of solifenacin was given for at least 40 weeks in the Fixed-dose assessment period. Children received solifenacin once daily during these 2 periods.
Period: Titration Period
Arm/Group | Solifenacin Succinate
Started | 23
Treated | 23
Completed | 22
Not Completed | 1
Not completed — Protocol Deviation | 1
Period: Fixed-Dose Assessment Period
Arm/Group | Solifenacin Succinate
Started | 22
Treated | 22
Completed | 21
Not Completed | 1
Not completed — Lack of Efficacy | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set (SAF), which consisted of all participants who took at least one dose of study drug. For the MCC baseline characteristic: Full Analysis Set (FAS), which consisted of all participants who took at least one dose of study drug and provided both valid baseline and at least one post-baseline value for primary endpoint.
Arm/Group | Solifenacin Succinate
Number analyzed (Participants) | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 23
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: months] | 35.3 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 9
Weight [Mean (Standard Deviation); unit: kg] | 13.2 (2.87)
Duration of NDO Disease [Median (Full Range); unit: years] — Population: SAF population
  years | 1.99 [0.13 to 4.51]
Maximum Cystometric Capacity (MCC) [Mean (Standard Deviation); unit: mL] — Population: FAS population
  mL
    number analyzed (Participants) | 21
    (all) | 92.3 (38.2)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 24 in Maximum Cystometric Capacity (MCC)
Description: MCC was the volume instilled into the bladder prior to leakage or end of bladder-filling (whichever was reached first), as assessed by urodynamics (procedure: the bladder was to be filled until voiding/leakage began, or until it was stopped because either the participant experienced pain or discomfort or 135% of expected bladder capacity [EBC] was reached for participants ≥ 2 years or of maximum catheterized volume [MCV] for participants aged 6 months to < 2 years; the participants' bladder was emptied via catheterization).
Time Frame: Baseline and Week 24
Population: Full Analysis Set (FAS), which consisted of all participants who took at least one dose of study drug and provided both valid baseline and at least one post-baseline value for the primary efficacy endpoint.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Solifenacin Succinate
Number analyzed (Participants) | 21
mL | 37.0 (35.9)
Statistical Analysis 1: Comparison: Solifenacin Succinate; Week 24 MCC Analysis; Test type: Other; p < 0.001, t-test, 2 sided — From a 2-sided one sample t-test, testing the null hypothesis that change from baseline = 0

2. Secondary Outcome: Change From Baseline to Weeks 3, 6, 9, 12 and 52 in MCC
Description: MCC was the volume instilled into the bladder prior to leakage or end of bladder-filling (whichever was reached first) as assessed by urodynamics (procedure: the bladder was to be filled until voiding/leakage began, or until it was stopped because either the participant experienced pain or discomfort or 135% of EBC was reached for participants ≥ 2 years or of MCV for participants aged 6 months to < 2 years. The participants' bladder was emptied via catheterization).
Time Frame: Baseline and Weeks 3, 6, 9, 12, 52
Population: FAS population with available data at baseline and at each time point.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Solifenacin Succinate
Number analyzed (Participants) | 21
mL
  Week 3: number analyzed (Participants) | 11
  Week 3 | 45.2 (44.8)
  Week 6: number analyzed (Participants) | 11
  Week 6 | 36.5 (36.6)
  Week 9: number analyzed (Participants) | 8
  Week 9 | 23.9 (57.6)
  Week 12: number analyzed (Participants) | 16
  Week 12 | 40.2 (37.9)
  Week 52: number analyzed (Participants) | 14
  Week 52 | 58.6 (34.1)

3. Secondary Outcome: Change From Baseline to Weeks 3, 6, 9, 12, 24 and 52 in Bladder Compliance
Description: Bladder compliance gives an indication of the elasticity of the bladder wall. Bladder compliance was calculated by dividing the change in volume during the filling of the bladder by the change in detrusor pressure during that change in bladder volume using urodynamic assessments. The values for bladder volume and detrusor pressure at the beginning and end of filling were taken and used.
Time Frame: Baseline and Weeks 3, 6, 9, 12, 24, 52
Population: FAS population with available data at baseline and at each time point.
Measure: Mean (Standard Deviation); unit: mL/cmH2O
Arm/Group | Solifenacin Succinate
Number analyzed (Participants) | 21
mL/cmH2O
  Week 3: number analyzed (Participants) | 11
  Week 3 | 4.55 (4.30)
  Week 6: number analyzed (Participants) | 11
  Week 6 | 5.45 (8.45)
  Week 9: number analyzed (Participants) | 8
  Week 9 | 10.00 (16.42)
  Week 12: number analyzed (Participants) | 16
  Week 12 | 4.14 (4.20)
  Week 24 | 5.10 (6.82)
  Week 52: number analyzed (Participants) | 14
  Week 52 | 5.94 (4.24)
Statistical Analysis 1: Comparison: Solifenacin Succinate; Week 24 Analysis; Test type: Other; p = 0.003, t-test, 2 sided — From a 2-sided one sample t-test, testing the null hypothesis that change from baseline=0

4. Secondary Outcome: Change From Baseline to Weeks 3, 6, 9, 12, 24 and 52 in Detrusor Pressure at End of Bladder-Filling
Description: Detrusor pressure was expressed as bladder pressure minus intra-abdominal pressure as assessed by urodynamics.
Time Frame: Baseline and Weeks 3, 6, 9, 12, 24, 52
Population: FAS population with available data at baseline and at each time point.
Measure: Mean (Standard Deviation); unit: cmH2O
Arm/Group | Solifenacin Succinate
Number analyzed (Participants) | 21
cmH2O
  Week 3: number analyzed (Participants) | 11
  Week 3 | -5.2 (12.9)
  Week 6: number analyzed (Participants) | 11
  Week 6 | -8.3 (14.8)
  Week 9: number analyzed (Participants) | 8
  Week 9 | -10.3 (18.2)
  Week 12: number analyzed (Participants) | 16
  Week 12 | -0.6 (23.4)
  Week 24 | -1.0 (13.9)
  Week 52: number analyzed (Participants) | 14
  Week 52 | -9.8 (19.2)
Statistical Analysis 1: Comparison: Solifenacin Succinate; Week 24 Analysis; Test type: Other; p = 0.744, t-test, 2 sided — From a 2-sided one sample t-test, testing the null hypothesis that change from baseline = 0

5. Secondary Outcome: Change From Baseline to Weeks 3, 6, 9, 12, 24 and 52 in Detrusor Pressure 5 Minutes After End of Bladder-Filling
Description: Detrusor pressure was expressed as bladder pressure minus intra-abdominal pressure as assessed by urodynamics.
Time Frame: Baseline and Weeks 3, 6, 9, 12, 24, 52
Population: FAS population with with available data at baseline and at each time point.
Measure: Mean (Standard Deviation); unit: cmH2O
Arm/Group | Solifenacin Succinate
Number analyzed (Participants) | 21
cmH2O
  Week 3: number analyzed (Participants) | 11
  Week 3 | 0.9 (8.4)
  Week 6: number analyzed (Participants) | 11
  Week 6 | 1.3 (10.4)
  Week 9: number analyzed (Participants) | 8
  Week 9 | 1.2 (11.8)
  Week 12: number analyzed (Participants) | 16
  Week 12 | -4.1 (10.9)
  Week 24 | -2.0 (9.4)
  Week 52: number analyzed (Participants) | 14
  Week 52 | -2.3 (14.7)
Statistical Analysis 1: Comparison: Solifenacin Succinate; Week 24 Analysis; Test type: Other; p = 0.352, t-test, 2 sided — From a 2-sided one sample t-test, testing the null hypothesis that change from baseline = 0

6. Secondary Outcome: Change From Baseline to Weeks 3, 6, 9, 12, 24 and 52 in Catheterized Volume 5 Minutes After End of Bladder-Filling
Description: Catheterized volume was measured when the bladder was emptied via catheterization 5 minutes after the end of bladder-filling.
Time Frame: Baseline and Weeks 3, 6, 9, 12, 24, 52
Population: FAS population with available data at baseline and at each time point.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Solifenacin Succinate
Number analyzed (Participants) | 15
mL
  Week 3: number analyzed (Participants) | 5
  Week 3 | 38.6 (52.6)
  Week 6: number analyzed (Participants) | 6
  Week 6 | 41.8 (25.5)
  Week 9: number analyzed (Participants) | 4
  Week 9 | 50.5 (40.5)
  Week 12: number analyzed (Participants) | 10
  Week 12 | 50.5 (46.6)
  Week 24: number analyzed (Participants) | 13
  Week 24 | 44.0 (29.5)
  Week 52: number analyzed (Participants) | 8
  Week 52 | 59.8 (27.0)
Statistical Analysis 1: Comparison: Solifenacin Succinate; Week 24 Analysis; Test type: Other; p < 0.001, t-test, 2 sided — From a 2-sided one sample t-test, testing the null hypothesis that change from baseline = 0

7. Secondary Outcome: Change From Baseline to Weeks 3, 6, 9, 12, 24 and 52 in Bladder Volume Until First Detrusor Contraction (> 15 cmH2O)
Description: Bladder volume as assessed by urodynamics.
Time Frame: Baseline and Weeks 3, 6, 9, 12, 24, 52
Population: FAS population with data available at baseline and at each time point and excluding participants who did not have a detrusor contraction.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Solifenacin Succinate
Number analyzed (Participants) | 21
mL
  Week 3: number analyzed (Participants) | 4
  Week 3 | 47.0 (31.3)
  Week 6: number analyzed (Participants) | 2
  Week 6 | 87.4 (57.4)
  Week 9: number analyzed (Participants) | 4
  Week 9 | 77.0 (86.2)
  Week 12: number analyzed (Participants) | 5
  Week 12 | 18.7 (37.5)
  Week 24: number analyzed (Participants) | 11
  Week 24 | 22.9 (52.3)
  Week 52: number analyzed (Participants) | 4
  Week 52 | 89.2 (58.0)
Statistical Analysis 1: Comparison: Solifenacin Succinate; Week 24 Analysis; Test type: Other; p = 0.177, t-test, 2 sided — From a 2-sided one sample t-test, testing the null hypothesis that change from baseline = 0

8. Secondary Outcome: Change From Baseline to Weeks 3, 6, 9, 12, 24 and 52 in Bladder Volume at 10 cmH20 Detrusor Pressure
Description: Bladder volume as assessed by urodynamics.
Time Frame: Baseline and Weeks 3, 6, 9, 12, 24, 52
Population: FAS population with data available at baseline and at each time point and whose pressure reached 10 cmH2O.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Solifenacin Succinate
Number analyzed (Participants) | 19
mL
  Week 3: number analyzed (Participants) | 8
  Week 3 | 31.9 (47.3)
  Week 6: number analyzed (Participants) | 8
  Week 6 | 47.8 (55.9)
  Week 9: number analyzed (Participants) | 6
  Week 9 | 31.5 (54.1)
  Week 12: number analyzed (Participants) | 14
  Week 12 | 30.1 (37.9)
  Week 24: number analyzed (Participants) | 17
  Week 24 | 28.7 (47.9)
  Week 52: number analyzed (Participants) | 10
  Week 52 | 49.4 (40.9)
Statistical Analysis 1: Comparison: Solifenacin Succinate; Week 24 Analyis; Test type: Other; p = 0.025, t-test, 2 sided — From a 2-sided one sample t-test, testing the null hypothesis that change from baseline = 0

9. Secondary Outcome: Change From Baseline to Weeks 3, 6, 9, 12, 24 and 52 in Bladder Volume at 20 cmH20 Detrusor Pressure
Description: Bladder volume as assessed by urodynamics.
Time Frame: Baseline and Weeks 3, 6, 9, 12, 24, 52
Population: FAS population with data available at baseline and at each time point and whose pressure reached 20 cmH2O.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Solifenacin Succinate
Number analyzed (Participants) | 13
mL
  Week 3: number analyzed (Participants) | 6
  Week 3 | 52.4 (59.4)
  Week 6: number analyzed (Participants) | 4
  Week 6 | 65.5 (54.9)
  Week 9: number analyzed (Participants) | 3
  Week 9 | 52.0 (58.0)
  Week 12: number analyzed (Participants) | 6
  Week 12 | 53.9 (67.6)
  Week 24: number analyzed (Participants) | 10
  Week 24 | 40.1 (56.2)
  Week 52: number analyzed (Participants) | 3
  Week 52 | 75.4 (71.6)
Statistical Analysis 1: Comparison: Solifenacin Succinate; Week 24 Analysis; Test type: Other; p = 0.050, t-test, 2 sided — From a 2-sided one sample t-test, testing the null hypothesis that change from baseline = 0

10. Secondary Outcome: Change From Baseline to Weeks 3, 6, 9, 12, 24 and 52 in Bladder Volume at 30 cmH20 Detrusor Pressure
Description: Bladder volume as assessed by urodynamics.
Time Frame: Baseline and Weeks 3, 6, 9, 12, 24, 52
Population: FAS population with data available at baseline and at each time point and whose pressure reached 30 cmH2O.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Solifenacin Succinate
Number analyzed (Participants) | 7
mL
  Week 3: number analyzed (Participants) | 2
  Week 3 | 101.9 (0.2)
  Week 6: number analyzed (Participants) | 1
  Week 6 | -2.3 (NA) — No data has been caluclated since data were only available for one participant.
  Week 9: number analyzed (Participants) | 2
  Week 9 | 76.0 (120.2)
  Week 12: number analyzed (Participants) | 2
  Week 12 | 74.7 (54.9)
  Week 24: number analyzed (Participants) | 2
  Week 24 | 67.5 (118.1)
  Week 52: number analyzed (Participants) | 1
  Week 52 | 93.6 (NA) — No data has been calculated since data were only available for one participant.
Statistical Analysis 1: Comparison: Solifenacin Succinate; Week 24 Analysis; Test type: Other; p = 0.567, t-test, 2 sided — From a 2-sided one sample t-test, testing the null hypothesis that change from baseline = 0

11. Secondary Outcome: Change From Baseline to Weeks 3, 6, 9, 12, 24 and 52 in Number of Overactive Detrusor Contractions (> 15 cmH2O) Until Leakage or End of Bladder-Filling
Time Frame: Baseline and Weeks 3, 6, 9, 12, 24, 52
Population: FAS population with data available at baseline and at each time point.
Measure: Mean (Standard Deviation); unit: contractions
Arm/Group | Solifenacin Succinate
Number analyzed (Participants) | 21
contractions
  Week 3: number analyzed (Participants) | 11
  Week 3 | -3.4 (3.9)
  Week 6: number analyzed (Participants) | 11
  Week 6 | -4.2 (5.3)
  Week 9: number analyzed (Participants) | 8
  Week 9 | -6.3 (6.6)
  Week 12: number analyzed (Participants) | 16
  Week 12 | -6.8 (8.9)
  Week 24 | -7.0 (8.6)
  Week 52: number analyzed (Participants) | 14
  Week 52 | -7.2 (10.2)
Statistical Analysis 1: Comparison: Solifenacin Succinate; Week 24 Analysis; Test type: Other; p = 0.001, t-test, 2 sided — From a 2-sided one sample t-test, testing the null hypothesis that change from baseline = 0

12. Secondary Outcome: Change From Baseline to Weeks 3, 6, 9, 12, 24, 36 and 52 in Average Catheterized Volume Per Catheterization
Description: The average catheterized volume per catheterization was calculated using all available (non-zero) catheterized volumes recorded over both of the 2 measuring days in the diary, whether or not these 2 days were concurrent. Catheterized volumes were recorded for 2 days in a participant diary prior to each visit. Four to six catheterizations were performed every day.
Time Frame: Baseline and Weeks 3, 6, 9, 12, 24, 36, 52
Population: FAS population with data available at baseline and at each time point.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Solifenacin Succinate
Number analyzed (Participants) | 18
mL
  Week 3 | 21.56 (26.16)
  Week 6: number analyzed (Participants) | 17
  Week 6 | 23.93 (23.80)
  Week 9 | 25.13 (24.91)
  Week 12 | 37.64 (22.43)
  Week 24 | 34.38 (33.04)
  Week 36: number analyzed (Participants) | 17
  Week 36 | 43.79 (34.13)
  Week 52: number analyzed (Participants) | 16
  Week 52 | 40.42 (31.83)
Statistical Analysis 1: Comparison: Solifenacin Succinate; Week 24 Analysis; Test type: Other; p < 0.001, t-test, 2 sided — From a 2-sided one sample t-test, testing the null hypothesis that change from baseline = 0

13. Secondary Outcome: Change From Baseline to Weeks 3, 6, 9, 12, 24, 36 and 52 in Maximum Catheterized Volume (MCV)
Description: The maximum catheterized volume per day was calculated using all available (non-zero) catheterized volumes recorded for the 2 measuring days in the diary, whether or not these 2 days were concurrent. The maximum value was calculated separately for each measuring day and the mean of these two values was used.
Time Frame: Baseline and Weeks 3, 6, 9, 12, 24, 36, 52
Population: FAS population with data available at baseline and at each time point.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Solifenacin Succinate
Number analyzed (Participants) | 18
mL
  Week 3 | 30.00 (32.06)
  Week 6: number analyzed (Participants) | 17
  Week 6 | 31.06 (34.36)
  Week 9 | 27.31 (33.34)
  Week 12 | 40.56 (24.64)
  Week 24 | 40.56 (51.45)
  Week 36: number analyzed (Participants) | 17
  Week 36 | 57.91 (47.67)
  Week 52: number analyzed (Participants) | 16
  Week 52 | 41.69 (46.71)
Statistical Analysis 1: Comparison: Solifenacin Succinate; Week 24 Analysis; Test type: Other; p = 0.004, t-test, 2 sided — From a 2-sided one sample t-test, testing the null hypothesis that change from baseline = 0

14. Secondary Outcome: Change From Baseline to Weeks 3, 6, 9, 12, 24, 36 and 52 in Average First Morning Catheterized Volume
Description: The first morning catheterized volume was the volume associated with the first morning catheterization. The average first morning catheterized volume was calculated as the average of the available first morning catheterized volumes recorded for the 2 measuring days in the diary, whether or not these 2 days are concurrent.
Time Frame: Baseline and Weeks 3, 6, 9, 12, 24, 36, 52
Population: FAS population with data available at baseline and at each time point.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Solifenacin Succinate
Number analyzed (Participants) | 18
mL
  Week 3 | 19.47 (34.74)
  Week 6: number analyzed (Participants) | 17
  Week 6 | 24.26 (35.49)
  Week 9 | 23.06 (36.50)
  Week 12 | 32.56 (35.97)
  Week 24 | 40.58 (41.89)
  Week 36: number analyzed (Participants) | 17
  Week 36 | 40.62 (44.14)
  Week 52: number analyzed (Participants) | 16
  Week 52 | 39.88 (34.91)
Statistical Analysis 1: Comparison: Solifenacin Succinate; Week 24 Analysis; Test type: Other; p = 0.001, t-test, 2 sided — From a 2-sided one sample t-test, testing the null hypothesis that change from baseline = 0

15. Secondary Outcome: Change From Baseline to Weeks 3, 6, 9, 12, 24, 36 and 52 in Mean Number of Periods Between the Clean Intermittent Catheterizations (CICs) With Incontinence Per 24 Hours
Description: Participants were required to have 4-6 CICs per day on a schedule fixed for the duration of the study. To calculate the number of periods between CICs with incontinence in a diary day, the diary day was divided into periods between CICs (i.e. inter-CIC periods). The hour period, rather than the exact time, of each CIC and incontinence episode was recorded in the diary. When an incontinence episode and a CIC were marked in the same hour period, the incontinence episode was counted as occurring prior to the CIC (when the bladder had not yet emptied), rather than after it (when the bladder had recently been emptied), i.e. the inter-CIC period ended with the hour in which the CIC was recorded. The mean number of periods between CICs with incontinence per 24 hours was the number of periods between CICs when incontinence occurred, divided by the total number of valid diary days.
Time Frame: Baseline and Weeks 3, 6, 9, 12, 24, 36, 52
Population: FAS population with data available at baseline and at each time point.
Measure: Mean (Standard Deviation); unit: periods
Arm/Group | Solifenacin Succinate
Number analyzed (Participants) | 17
periods
  Week 3 | -1.18 (1.42)
  Week 6: number analyzed (Participants) | 15
  Week 6 | -1.38 (1.21)
  Week 9: number analyzed (Participants) | 15
  Week 9 | -1.47 (1.19)
  Week 12: number analyzed (Participants) | 16
  Week 12 | -1.25 (1.32)
  Week 24 | -1.31 (1.39)
  Week 36: number analyzed (Participants) | 16
  Week 36 | -1.06 (1.25)
  Week 52: number analyzed (Participants) | 14
  Week 52 | -1.29 (1.42)
Statistical Analysis 1: Comparison: Solifenacin Succinate; Week 24 Analysis; Test type: Other; p = 0.001, t-test, 2 sided — From a 2-sided one sample t-test, testing the null hypothesis that change from baseline = 0

16. Secondary Outcome: Percentage of Days With Catheterizations for Each Hour of 24 Hour Day at Baseline
Description: For each one hour period of the 24 hour day, the percentage of days with catheterization was assessed as the number of days with catheterization occurring within the one hour period divided by the number of valid diary days over all participants. Each participant contributed to up to three days of valid diary data for each visit.
Time Frame: 3 days prior to Baseline visit
Population: FAS population.
Measure: Number; unit: percentage of days with catheterization
Units Other Than Participants: Days
Arm/Group | Solifenacin Succinate
Number analyzed (Participants) | 21
Number analyzed (Days) | 54
percentage of days with catheterization
  06:00-07:00 | 46.3
  07:00-08:00 | 29.6
  08:00-09:00 | 18.5
  09:00-10:00 | 27.8
  10:00-11:00 | 16.7
  11:00-12:00 | 22.2
  12:00-13:00 | 44.4
  13:00-14:00 | 20.4
  14:00-15:00 | 20.4
  15:00-16:00 | 24.1
  16:00-17:00 | 27.8
  17:00-18:00 | 14.8
  18:00-19:00 | 40.7
  19:00-20:00 | 31.5
  20:00-21:00 | 13.0
  21:00-22:00 | 38.9
  22:00-23:00 | 14.8
  23:00-00:00 | 13.0
  00:00-01:00 | 24.1
  01:00-02:00 | 9.3
  02:00-03:00 | 1.9
  03:00-04:00 | 3.7
  04:00-05:00 | 0
  05:00-06:00 | 13.0

17. Secondary Outcome: Percentage of Days With Catheterizations for Each Hour of 24 Hour Day During Week 3
Description: as for outcome 16
Time Frame: 3 days prior to Week 3 visit
Population: FAS population.
Measure: Number; unit: percentage of days with catheterization
Units Other Than Participants: Days
Arm/Group | Solifenacin Succinate
Number analyzed (Participants) | 21
Number analyzed (Days) | 63
percentage of days with catheterization
  06:00-07:00 | 36.5
  07:00-08:00 | 30.2
  08:00-09:00 | 20.6
  09:00-10:00 | 27.0
  10:00-11:00 | 20.6
  11:00-12:00 | 19.0
  12:00-13:00 | 36.5
  13:00-14:00 | 34.9
  14:00-15:00 | 15.9
  15:00-16:00 | 23.8
  16:00-17:00 | 20.6
  17:00-18:00 | 28.6
  18:00-19:00 | 36.5
  19:00-20:00 | 25.4
  20:00-21:00 | 20.6
  21:00-22:00 | 36.5
  22:00-23:00 | 17.5
  23:00-00:00 | 9.5
  00:00-01:00 | 25.4
  01:00-02:00 | 12.7
  02:00-03:00 | 3.2
  03:00-04:00 | 0
  04:00-05:00 | 0
  05:00-06:00 | 11.1

18. Secondary Outcome: Percentage of Days With Catheterizations for Each Hour of 24 Hour Day During Week 6
Description: as for outcome 16
Time Frame: 3 days prior to Week 6 visit
Population: FAS population.
Measure: Number; unit: percentage of days with catheterization
Units Other Than Participants: Days
Arm/Group | Solifenacin Succinate
Number analyzed (Participants) | 21
Number analyzed (Days) | 60
percentage of days with catheterization
  06:00-07:00 | 35.0
  07:00-08:00 | 30.0
  08:00-09:00 | 20.0
  09:00-10:00 | 36.7
  10:00-11:00 | 15.0
  11:00-12:00 | 11.7
  12:00-13:00 | 43.3
  13:00-14:00 | 33.3
  14:00-15:00 | 15.0
  15:00-16:00 | 30.0
  16:00-17:00 | 25.0
  17:00-18:00 | 20.0
  18:00-19:00 | 35.0
  19:00-20:00 | 28.3
  20:00-21:00 | 11.7
  21:00-22:00 | 40.0
  22:00-23:00 | 18.3
  23:00-00:00 | 16.7
  00:00-01:00 | 18.3
  01:00-02:00 | 0
  02:00-03:00 | 5.0
  03:00-04:00 | 3.3
  04:00-05:00 | 0
  05:00-06:00 | 6.7

19. Secondary Outcome: Percentage of Days With Catheterizations for Each Hour of 24 Hour Day During Week 9
Description: as for outcome 16
Time Frame: 3 days prior to Week 9 visit
Population: FAS population.
Measure: Number; unit: percentage of days with catheterization
Units Other Than Participants: Days
Arm/Group | Solifenacin Succinate
Number analyzed (Participants) | 21
Number analyzed (Days) | 63
percentage of days with catheterization
  06:00-07:00 | 34.9
  07:00-08:00 | 36.5
  08:00-09:00 | 19.0
  09:00-10:00 | 23.8
  10:00-11:00 | 17.5
  11:00-12:00 | 19.0
  12:00-13:00 | 42.9
  13:00-14:00 | 27.0
  14:00-15:00 | 17.5
  15:00-16:00 | 31.7
  16:00-17:00 | 15.9
  17:00-18:00 | 23.8
  18:00-19:00 | 38.1
  19:00-20:00 | 27.0
  20:00-21:00 | 17.5
  21:00-22:00 | 38.1
  22:00-23:00 | 12.7
  23:00-00:00 | 19.0
  00:00-01:00 | 19.0
  01:00-02:00 | 4.8
  02:00-03:00 | 1.6
  03:00-04:00 | 1.6
  04:00-05:00 | 1.6
  05:00-06:00 | 9.5

20. Secondary Outcome: Percentage of Days With Catheterizations for Each Hour of 24 Hour Day During Week 12
Description: as for outcome 16
Time Frame: 3 days prior to Week 12 visit
Population: FAS population.
Measure: Number; unit: percentage of days with catheterization
Units Other Than Participants: Days
Arm/Group | Solifenacin Succinate
Number analyzed (Participants) | 21
Number analyzed (Days) | 63
percentage of days with catheterization
  06:00-07:00 | 39.7
  07:00-08:00 | 31.7
  08:00-09:00 | 20.6
  09:00-10:00 | 27.0
  10:00-11:00 | 19.0
  11:00-12:00 | 15.9
  12:00-13:00 | 58.7
  13:00-14:00 | 19.0
  14:00-15:00 | 12.7
  15:00-16:00 | 22.2
  16:00-17:00 | 31.7
  17:00-18:00 | 15.9
  18:00-19:00 | 41.3
  19:00-20:00 | 22.2
  20:00-21:00 | 27.0
  21:00-22:00 | 38.1
  22:00-23:00 | 11.1
  23:00-00:00 | 14.3
  00:00-01:00 | 30.2
  01:00-02:00 | 1.6
  02:00-03:00 | 3.2
  03:00-04:00 | 3.2
  04:00-05:00 | 0
  05:00-06:00 | 6.3

21. Secondary Outcome: Percentage of Days With Catheterizations for Each Hour of 24 Hour Day During Week 24
Description: as for outcome 16
Time Frame: 3 days prior to Week 24 visit
Population: FAS population.
Measure: Number; unit: percentage of days with catheterization
Units Other Than Participants: Days
Arm/Group | Solifenacin Succinate
Number analyzed (Participants) | 21
Number analyzed (Days) | 63
percentage of days with catheterization
  06:00-07:00 | 33.3
  07:00-08:00 | 33.3
  08:00-09:00 | 22.2
  09:00-10:00 | 15.9
  10:00-11:00 | 23.8
  11:00-12:00 | 19.0
  12:00-13:00 | 44.4
  13:00-14:00 | 33.3
  14:00-15:00 | 9.5
  15:00-16:00 | 23.8
  16:00-17:00 | 27.0
  17:00-18:00 | 27.0
  18:00-19:00 | 34.9
  19:00-20:00 | 30.2
  20:00-21:00 | 20.6
  21:00-22:00 | 38.1
  22:00-23:00 | 6.3
  23:00-00:00 | 17.5
  00:00-01:00 | 25.4
  01:00-02:00 | 3.2
  02:00-03:00 | 3.2
  03:00-04:00 | 0
  04:00-05:00 | 0
  05:00-06:00 | 6.3

22. Secondary Outcome: Percentage of Days With Catheterizations for Each Hour of 24 Hour Day During Week 36
Description: as for outcome 16
Time Frame: 3 days prior to Week 36 visit
Population: FAS population.
Measure: Number; unit: percentage of days with catheterization
Units Other Than Participants: Days
Arm/Group | Solifenacin Succinate
Number analyzed (Participants) | 21
Number analyzed (Days) | 60
percentage of days with catheterization
  06:00-07:00 | 36.7
  07:00-08:00 | 35.0
  08:00-09:00 | 26.7
  09:00-10:00 | 20.0
  10:00-11:00 | 16.7
  11:00-12:00 | 16.7
  12:00-13:00 | 53.3
  13:00-14:00 | 30.0
  14:00-15:00 | 8.3
  15:00-16:00 | 25.0
  16:00-17:00 | 26.7
  17:00-18:00 | 23.3
  18:00-19:00 | 43.3
  19:00-20:00 | 21.7
  20:00-21:00 | 23.3
  21:00-22:00 | 38.3
  22:00-23:00 | 5.0
  23:00-00:00 | 15.0
  00:00-01:00 | 25.0
  01:00-02:00 | 5.0
  02:00-03:00 | 1.7
  03:00-04:00 | 0
  04:00-05:00 | 1.7
  05:00-06:00 | 1.7

23. Secondary Outcome: Percentage of Days With Catheterizations for Each Hour of 24 Hour Day During Week 52
Description: For each one hour period of the 24 hour day, the percentage of days with catheterization was assessed as the number of days with catheterization occurring within the one hour period divided by the number of valid diary days over all subjects. Each participant contributed to up to three days of valid diary data for each visit.
Time Frame: 3 days prior to Week 52 visit
Population: FAS population.
Measure: Number; unit: percentage of days with catheterization
Units Other Than Participants: Days
Arm/Group | Solifenacin Succinate
Number analyzed (Participants) | 21
Number analyzed (Days) | 57
percentage of days with catheterization
  06:00-07:00 | 35.1
  07:00-08:00 | 33.3
  08:00-09:00 | 28.1
  09:00-10:00 | 22.8
  10:00-11:00 | 15.8
  11:00-12:00 | 17.5
  12:00-13:00 | 50.9
  13:00-14:00 | 26.3
  14:00-15:00 | 10.5
  15:00-16:00 | 28.1
  16:00-17:00 | 19.3
  17:00-18:00 | 24.6
  18:00-19:00 | 45.6
  19:00-20:00 | 24.6
  20:00-21:00 | 21.1
  21:00-22:00 | 36.8
  22:00-23:00 | 15.8
  23:00-00:00 | 19.3
  00:00-01:00 | 14.0
  01:00-02:00 | 0
  02:00-03:00 | 0
  03:00-04:00 | 0
  04:00-05:00 | 0
  05:00-06:00 | 3.5

24. Secondary Outcome: Percentage of Days With Incontinence for Each Hour of 24 Hour Day at Baseline
Description: Incontinence was defined as leakage where a diaper is not used, or dampness where a diaper is used. For each one hour period of the 24 hour day, the percentage of days with incontinence was assessed as the number of days with incontinence occurring within the one hour period divided by the number of valid diary days over all participants. Each participant contributed to up to three days of valid diary data for each visit.
Time Frame: 3 days prior to Baseline visit
Population: FAS population.
Measure: Number; unit: percentage of days with incontinence
Units Other Than Participants: Days
Arm/Group | Solifenacin Succinate
Number analyzed (Participants) | 21
Number analyzed (Days) | 54
percentage of days with incontinence
  06:00-07:00 | 27.8
  07:00-08:00 | 27.8
  08:00-09:00 | 16.7
  09:00-10:00 | 37.0
  10:00-11:00 | 25.9
  11:00-12:00 | 22.2
  12:00-13:00 | 35.2
  13:00-14:00 | 33.3
  14:00-15:00 | 25.9
  15:00-16:00 | 31.5
  16:00-17:00 | 37.0
  17:00-18:00 | 24.1
  18:00-19:00 | 24.1
  19:00-20:00 | 31.5
  20:00-21:00 | 14.8
  21:00-22:00 | 35.2
  22:00-23:00 | 14.8
  23:00-00:00 | 9.3
  00:00-01:00 | 13.0
  01:00-02:00 | 5.6
  02:00-03:00 | 1.9
  03:00-04:00 | 1.9
  04:00-05:00 | 1.9
  05:00-06:00 | 7.4

25. Secondary Outcome: Percentage of Days With of Incontinence for Each Hour of 24 Hour Day During Week 3
Description: as for outcome 24
Time Frame: 3 days prior to Week 3 visit
Population: FAS population.
Measure: Number; unit: percentage of days with incontinence
Units Other Than Participants: Days
Arm/Group | Solifenacin Succinate
Number analyzed (Participants) | 21
Number analyzed (Days) | 63
percentage of days with incontinence
  06:00-07:00 | 17.5
  07:00-08:00 | 25.4
  08:00-09:00 | 11.1
  09:00-10:00 | 22.2
  10:00-11:00 | 22.2
  11:00-12:00 | 14.3
  12:00-13:00 | 15.9
  13:00-14:00 | 15.9
  14:00-15:00 | 20.6
  15:00-16:00 | 20.6
  16:00-17:00 | 15.9
  17:00-18:00 | 20.6
  18:00-19:00 | 14.3
  19:00-20:00 | 27.0
  20:00-21:00 | 19.0
  21:00-22:00 | 19.0
  22:00-23:00 | 3.2
  23:00-00:00 | 7.9
  00:00-01:00 | 4.8
  01:00-02:00 | 3.2
  02:00-03:00 | 1.6
  03:00-04:00 | 1.6
  04:00-05:00 | 0
  05:00-06:00 | 9.5

26. Secondary Outcome: Percentage of Days With Incontinence for Each Hour of 24 Hour Day During Week 6
Description: as for outcome 24
Time Frame: 3 days prior to Week 6 visit
Population: FAS population.
Measure: Number; unit: percentage of days with incontinence
Units Other Than Participants: Days
Arm/Group | Solifenacin Succinate
Number analyzed (Participants) | 21
Number analyzed (Days) | 60
percentage of days with incontinence
  06:00-07:00 | 25.0
  07:00-08:00 | 18.3
  08:00-09:00 | 11.7
  09:00-10:00 | 11.7
  10:00-11:00 | 20.0
  11:00-12:00 | 20.0
  12:00-13:00 | 13.3
  13:00-14:00 | 6.7
  14:00-15:00 | 11.7
  15:00-16:00 | 26.7
  16:00-17:00 | 21.7
  17:00-18:00 | 23.3
  18:00-19:00 | 15.0
  19:00-20:00 | 25.0
  20:00-21:00 | 10.0
  21:00-22:00 | 23.3
  22:00-23:00 | 5.0
  23:00-00:00 | 5.0
  00:00-01:00 | 0
  01:00-02:00 | 0
  02:00-03:00 | 3.3
  03:00-04:00 | 1.7
  04:00-05:00 | 3.3
  05:00-06:00 | 5.0

27. Secondary Outcome: Percentage of Days With Incontinence for Each Hour of 24 Hour Day During Week 9
Description: as for outcome 24
Time Frame: 3 days prior to Week 9 visit
Population: FAS population.
Measure: Number; unit: percentage of days with incontinence
Units Other Than Participants: Days
Arm/Group | Solifenacin Succinate
Number analyzed (Participants) | 21
Number analyzed (Days) | 63
percentage of days with incontinence
  06:00-07:00 | 14.3
  07:00-08:00 | 20.6
  08:00-09:00 | 9.5
  09:00-10:00 | 9.5
  10:00-11:00 | 25.4
  11:00-12:00 | 22.2
  12:00-13:00 | 11.1
  13:00-14:00 | 11.1
  14:00-15:00 | 12.7
  15:00-16:00 | 22.2
  16:00-17:00 | 20.6
  17:00-18:00 | 20.6
  18:00-19:00 | 11.1
  19:00-20:00 | 15.9
  20:00-21:00 | 14.3
  21:00-22:00 | 11.1
  22:00-23:00 | 6.3
  23:00-00:00 | 4.8
  00:00-01:00 | 1.6
  01:00-02:00 | 3.2
  02:00-03:00 | 1.6
  03:00-04:00 | 3.2
  04:00-05:00 | 1.6
  05:00-06:00 | 9.5

28. Secondary Outcome: Percentage of Days With Incontinence for Each Hour of 24 Hour Day During Week 12
Description: as for outcome 24
Time Frame: 3 days prior to Week 12 visit
Population: FAS population
Measure: Number; unit: percentage of days with incontinence
Units Other Than Participants: Days
Arm/Group | Solifenacin Succinate
Number analyzed (Participants) | 21
Number analyzed (Days) | 63
percentage of days with incontinence
  06:00-07:00 | 17.5
  07:00-08:00 | 11.1
  08:00-09:00 | 9.5
  09:00-10:00 | 28.6
  10:00-11:00 | 22.2
  11:00-12:00 | 23.8
  12:00-13:00 | 25.4
  13:00-14:00 | 4.8
  14:00-15:00 | 9.5
  15:00-16:00 | 28.6
  16:00-17:00 | 12.7
  17:00-18:00 | 17.5
  18:00-19:00 | 17.5
  19:00-20:00 | 17.5
  20:00-21:00 | 12.7
  21:00-22:00 | 11.1
  22:00-23:00 | 9.5
  23:00-00:00 | 6.3
  00:00-01:00 | 4.8
  01:00-02:00 | 1.6
  02:00-03:00 | 1.6
  03:00-04:00 | 1.6
  04:00-05:00 | 0
  05:00-06:00 | 7.9

29. Secondary Outcome: Percentage of Days With Incontinence for Each Hour of 24 Hour Day During Week 24
Description: as for outcome 24
Time Frame: 3 days prior to Week 24 visit
Population: FAS population.
Measure: Number; unit: percentage of days with incontinence
Units Other Than Participants: Days
Arm/Group | Solifenacin Succinate
Number analyzed (Participants) | 21
Number analyzed (Days) | 63
percentage of days with incontinence
  06:00-07:00 | 25.4
  07:00-08:00 | 14.3
  08:00-09:00 | 7.9
  09:00-10:00 | 15.9
  10:00-11:00 | 31.7
  11:00-12:00 | 23.8
  12:00-13:00 | 11.1
  13:00-14:00 | 11.1
  14:00-15:00 | 9.5
  15:00-16:00 | 25.4
  16:00-17:00 | 14.3
  17:00-18:00 | 30.2
  18:00-19:00 | 17.5
  19:00-20:00 | 19.0
  20:00-21:00 | 15.9
  21:00-22:00 | 7.9
  22:00-23:00 | 7.9
  23:00-00:00 | 6.3
  00:00-01:00 | 3.2
  01:00-02:00 | 3.2
  02:00-03:00 | 1.6
  03:00-04:00 | 0
  04:00-05:00 | 0
  05:00-06:00 | 4.8

30. Secondary Outcome: Percentage of Days With Incontinence for Each Hour of 24 Hour Day During Week 36
Description: as for outcome 24
Time Frame: 3 days prior to Week 36 visit
Population: FAS population.
Measure: Number; unit: percentage of days with incontinence
Units Other Than Participants: Days
Arm/Group | Solifenacin Succinate
Number analyzed (Participants) | 21
Number analyzed (Days) | 60
percentage of days with incontinence
  06:00-07:00 | 25.0
  07:00-08:00 | 13.3
  08:00-09:00 | 11.7
  09:00-10:00 | 18.3
  10:00-11:00 | 20.0
  11:00-12:00 | 20.0
  12:00-13:00 | 21.7
  13:00-14:00 | 13.3
  14:00-15:00 | 11.7
  15:00-16:00 | 31.7
  16:00-17:00 | 11.7
  17:00-18:00 | 16.7
  18:00-19:00 | 11.7
  19:00-20:00 | 30.0
  20:00-21:00 | 21.7
  21:00-22:00 | 18.3
  22:00-23:00 | 5.0
  23:00-00:00 | 11.7
  00:00-01:00 | 6.7
  01:00-02:00 | 3.3
  02:00-03:00 | 0
  03:00-04:00 | 1.7
  04:00-05:00 | 1.7
  05:00-06:00 | 5.0

31. Secondary Outcome: Percentage of Days With Incontinence for Each Hour of 24 Hour Day During Week 52
Description: as for outcome 24
Time Frame: 3 days prior to Week 52 visit
Population: FAS population.
Measure: Number; unit: percentage of days with incontinence
Units Other Than Participants: Days
Arm/Group | Solifenacin Succinate
Number analyzed (Participants) | 21
Number analyzed (Days) | 57
percentage of days with incontinence
  06:00-07:00 | 19.3
  07:00-08:00 | 19.3
  08:00-09:00 | 17.5
  09:00-10:00 | 14.0
  10:00-11:00 | 24.6
  11:00-12:00 | 33.3
  12:00-13:00 | 17.5
  13:00-14:00 | 8.8
  14:00-15:00 | 12.3
  15:00-16:00 | 29.8
  16:00-17:00 | 17.5
  17:00-18:00 | 22.8
  18:00-19:00 | 19.3
  19:00-20:00 | 21.1
  20:00-21:00 | 17.5
  21:00-22:00 | 21.1
  22:00-23:00 | 1.8
  23:00-00:00 | 3.5
  00:00-01:00 | 5.3
  01:00-02:00 | 3.5
  02:00-03:00 | 3.5
  03:00-04:00 | 1.8
  04:00-05:00 | 5.3
  05:00-06:00 | 3.5

32. Secondary Outcome: Change From Baseline to Week 24 and 52 in Infant and Toddler Quality of Life Short Form-47 Questionnaire (ITQoL SF-47) - Overall Health Score
Description: The ITQoL SF-47 consisted of 47 individual items and was filled in by the child's parent. The individual items are based on Likert scales with either 5 responses (coded as 1 through to 5) or 4 responses (coded as 1 through to 4). From subsets of these coded values, 11 scales are derived: overall health, physical activities, development, discomfort, moods and temperaments, perceptions of current past and future health and perception of changes. Each scale score ranges from 0 (worst possible) to 100 (best possible).
Time Frame: Baseline and Weeks 24, 52
Population: FAS population with available data at baseline and at each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Solifenacin Succinate
Number analyzed (Participants) | 20
units on a scale
  Week 24 | -1.8 (19.2)
  Week 52: number analyzed (Participants) | 15
  Week 52 | 9.0 (17.4)
Statistical Analysis 1: Comparison: Solifenacin Succinate; Week 24 Analysis; Test type: Other; p = 0.688, t-test, 2 sided — From a 2-sided one sample t-test, testing the null hypothesis that change from baseline = 0

33. Secondary Outcome: Change From Baseline to Week 24 and 52 in ITQoL SF-47 - Physical Abilities Score
Description: as for outcome 32
Time Frame: Baseline and Weeks 24, 52
Population: FAS population with data available at baseline and at each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Solifenacin Succinate
Number analyzed (Participants) | 20
units on a scale
  Week 24 | 2.17 (18.70)
  Week 52: number analyzed (Participants) | 15
  Week 52 | 3.93 (14.81)
Statistical Analysis 1: Comparison: Solifenacin Succinate; Week 24 Analysis; Test type: Other; p = 0.610, t-test, 2 sided — From a 2-sided one sample t-test, testing the null hypothesis that change from baseline = 0

34. Secondary Outcome: Change From Baseline to Week 24 and 52 in ITQoL SF-47 - Growth and Development Score
Description: as for outcome 32
Time Frame: Baseline and Weeks 24, 52
Population: FAS population with data available at baseline and at each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Solifenacin Succinate
Number analyzed (Participants) | 20
units on a scale
  Week 24 | -1.50 (11.37)
  Week 52: number analyzed (Participants) | 15
  Week 52 | 2.33 (13.21)
Statistical Analysis 1: Comparison: Solifenacin Succinate; Week 24 Analysis; Test type: Other; p = 0.562, t-test, 2 sided — From a 2-sided one sample t-test, testing the null hypothesis that change from baseline = 0

35. Secondary Outcome: Change From Baseline to Week 24 and 52 in ITQoL SF-47 - Pain Score
Description: as for outcome 32
Time Frame: Baseline and Weeks 24, 52
Population: FAS population with data available at baseline and at each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Solifenacin Succinate
Number analyzed (Participants) | 19
units on a scale
  Week 24: number analyzed (Participants) | 18
  Week 24 | -3.47 (32.60)
  Week 52: number analyzed (Participants) | 15
  Week 52 | -0.83 (21.37)
Statistical Analysis 1: Comparison: Solifenacin Succinate; Week 24 Analysis; Test type: Other; p = 0.657, t-test, 2 sided — From a 2-sided one sample t-test, testing the null hypothesis that change from baseline = 0

36. Secondary Outcome: Change From Baseline to Week 24 and 52 in ITQoL SF-47 - Temperament and Moods Score
Description: as for outcome 32
Time Frame: Baseline and Weeks 24, 52
Population: FAS population with data available at baseline and at each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Solifenacin Succinate
Number analyzed (Participants) | 19
units on a scale
  Week 24: number analyzed (Participants) | 18
  Week 24 | -1.85 (16.06)
  Week 52: number analyzed (Participants) | 15
  Week 52 | -1.11 (16.02)
Statistical Analysis 1: Comparison: Solifenacin Succinate; Week 24 Analysis; Test type: Other; p = 0.631, t-test, 2 sided — From a 2-sided one sample t-test, testing the null hypothesis that change from baseline = 0

37. Secondary Outcome: Change From Baseline to Week 24 and 52 in ITQoL SF-47 - Behaviour Score
Description: as for outcome 32
Time Frame: Baseline and Weeks 24, 52
Population: FAS population with data available at baseline and at each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Solifenacin Succinate
Number analyzed (Participants) | 18
units on a scale
  Week 24: number analyzed (Participants) | 17
  Week 24 | -1.69 (8.24)
  Week 52: number analyzed (Participants) | 13
  Week 52 | -0.06 (6.86)
Statistical Analysis 1: Comparison: Solifenacin Succinate; Week 24 Analysis; Test type: Other; p = 0.410, t-test, 2 sided — From a 2-sided one sample t-test, testing the null hypothesis that change from baseline = 0

38. Secondary Outcome: Change From Baseline to Week 24 and 52 in ITQoL SF-47 - General Health Score
Description: as for outcome 32
Time Frame: Baseline and Weeks 24, 52
Population: FAS population with data available at baseline and at each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Solifenacin Succinate
Number analyzed (Participants) | 18
units on a scale
  Week 24: number analyzed (Participants) | 17
  Week 24 | 0.39 (21.16)
  Week 52: number analyzed (Participants) | 13
  Week 52 | 4.29 (17.39)
Statistical Analysis 1: Comparison: Solifenacin Succinate; Week 24 Analysis; Test type: Other; p = 0.940, t-test, 2 sided — From a 2-sided one sample t-test, testing the null hypothesis that change from baseline = 0

39. Secondary Outcome: Change From Baseline to Week 24 and 52 in ITQoL SF-47 - Change in Health Score
Description: as for outcome 32
Time Frame: Baseline and Weeks 24, 52
Population: FAS population with data available at baseline and at each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Solifenacin Succinate
Number analyzed (Participants) | 18
units on a scale
  Week 24: number analyzed (Participants) | 17
  Week 24 | 0.00 (23.39)
  Week 52: number analyzed (Participants) | 13
  Week 52 | 5.77 (20.80)
Statistical Analysis 1: Comparison: Solifenacin Succinate; Week 24 Analysis; Test type: Other; p = 1.000, t-test, 2 sided — From a 2-sided one sample t-test, testing the null hypothesis that change from baseline = 0

40. Secondary Outcome: Change From Baseline to Week 24 and 52 in ITQoL SF-47 - Parent-Emotional Impact Score
Description: as for outcome 32
Time Frame: Baseline and Weeks 24, 52
Population: FAS population with data available at baseline and at each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Solifenacin Succinate
Number analyzed (Participants) | 18
units on a scale
  Week 24: number analyzed (Participants) | 17
  Week 24 | -3.31 (23.81)
  Week 52: number analyzed (Participants) | 13
  Week 52 | 4.81 (28.20)
Statistical Analysis 1: Comparison: Solifenacin Succinate; Week 24 Analysis; Test type: Other; p = 0.575, t-test, 2 sided — From a 2-sided one sample t-test, testing the null hypothesis that change from baseline = 0

41. Secondary Outcome: Change From Baseline to Week 24 and 52 in ITQoL SF-47 - Parent-Time Impact Score
Description: as for outcome 32
Time Frame: Baseline and Weeks 24, 52
Population: FAS population with data available at baseline and at each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Solifenacin Succinate
Number analyzed (Participants) | 18
units on a scale
  Week 24: number analyzed (Participants) | 17
  Week 24 | 15.2 (26.6)
  Week 52: number analyzed (Participants) | 13
  Week 52 | 7.1 (24.5)
Statistical Analysis 1: Comparison: Solifenacin Succinate; Week 24 Analysis; Test type: Other; p = 0.031, t-test, 2 sided — From a 2-sided one sample t-test, testing the null hypothesis that change from baseline = 0

42. Secondary Outcome: Change From Baseline to Week 24 and 52 in ITQoL SF-47 - Family Cohesion Impact Score
Description: as for outcome 32
Time Frame: Baseline and Weeks 24, 52
Population: FAS population with data available at baseline and at each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Solifenacin Succinate
Number analyzed (Participants) | 18
units on a scale
  Week 24: number analyzed (Participants) | 17
  Week 24 | 1.5 (16.7)
  Week 52: number analyzed (Participants) | 13
  Week 52 | -4.2 (17.7)
Statistical Analysis 1: Comparison: Solifenacin Succinate; Week 24 Analysis; Test type: Other; p = 0.721, t-test, 2 sided — From a 2-sided one sample t-test, testing the null hypothesis that change from baseline = 0

ADVERSE EVENTS:
Time Frame: From first dose of study drug to last dose of study drug (up to 54 weeks)
Arm/Group | Solifenacin Succinate
All-Cause Mortality (participants affected / at risk) | 0/23
Serious Adverse Events (participants affected / at risk) | 3/23
Other Adverse Events (participants affected / at risk) | 11/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Solifenacin Succinate (N=23)
Teratoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Vomiting (Gastrointestinal disorders) | 1
Pharyngitis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Solifenacin Succinate (N=23)
Constipation (Gastrointestinal disorders) | 3
Dental caries (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Dry mouth (Gastrointestinal disorders) | 2
Enteritis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Pyrexia (General disorders) | 1
Bronchitis (Infections and infestations) | 1
Escherichia urinary tract infection (Infections and infestations) | 2
Gastroenteritis (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 4
Otitis media (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 1
Tonsillitis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 3
Urinary tract infection (Infections and infestations) | 2
Urinary tract infection bacterial (Infections and infestations) | 3
Urinary tract infection enterococcal (Infections and infestations) | 1
Burns second degree (Injury, poisoning and procedural complications) | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1
Bacterial test positive (Investigations) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data. Sponsor must receive a site's manuscript sixty (60) days prior to publication for review and comment.